CLINICAL TRIAL: NCT01616823
Title: Duration of Rupture of Membranes and Risk of Fetal Transmission of HIV in Optimally Managed HIV Positive Mothers
Brief Title: Fetal HIV Transmission Risk and Duration of Membrane Rupture
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 10-232
Record Dates: First submitted 2012-02-29; First posted 2012-06-12 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Human Immunodeficiency Virus; HIV
Keywords: Human immunodeficiency virus (HIV) positive women
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV Positive Women: HIV positive women in two downtown Toronto, Ontario academic-affiliated hospitals

SUMMARY:
In optimally managed HIV+ women with undetectable viral loads, who are on HAART and also receiving intrapartum IV ZDV, the risk of vertical transmission of HIV is independent of the length of time of rupture of membranes.

DETAILED DESCRIPTION:
In developed countries, HIV infection is now considered a chronic disease and thus the life expectancy of people infected with HIV is approaching that of the general population. Therefore many HIV positive women are choosing to pursue pregnancies. An important concern for antenatal and intrapartum management is decreasing the risk of vertical transmission. With the use of highly active antiretroviral therapy (HAART) and intrapartum IV zidovudine (ZDV) the risk of transmission is decreased significantly, however there is some debate surrounding optimal mode of delivery. Possible mechanisms leading to perinatal transmission include transfusion of the mother's blood to the fetus during labour contractions, infection after rupture of membranes and direct contact of the fetus with infected secretions or blood from the maternal genital tract.

When maternal viral load is detectable, The Society of Obstetricians and Gynaecologists of Canada (SOGC) and other governing bodies recommend that elective cesarean section be performed for delivery as there is a 12-fold increased risk of perinatal transmission. However, the evidence suggests that for women at very low risk of transmission, such as those with an undetectable viral load and on HAART, the benefit of transmission reduction provided by cesarean section may be negligible.

The question of length of time of rupture of membranes prior to delivery and transmission risk has been a source of controversy, especially in the context of women on suppressive therapy (HAART) with an undetectable viral load. Traditional thinking has stated that the length of time of rupture of membranes should not be longer than 4 hours, as the benefit of cesarean section is lost after this time. However, this thinking is based on data where maternal viral loads were not known and only intrapartum IV ZDV was used. Many practitioners believe that in women with undetectable viral loads, virally suppressed on HAART, the safest route of delivery is vaginal, irrespective of length of time of rupture of membranes.

This is a retrospective cohort study which plans to examine the mode of delivery and median length of time of rupture of membranes for HIV positive women in two downtown academic institutions in Toronto.

ELIGIBILITY:
Inclusion Criteria:

* all HIV positive women from January 2000

Exclusion Criteria:

* women not on HAART and who were not receiving intrapartum intravenous zidovudine

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Total of 210 women from two downtown Toronto, Ontario academic-affiliated hospitals
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Mode of delivery | Ten years
  In optimally managed HIV+ women with undetectable viral loads and on HAART, receiving intrapartum IV ZDV, the risk of vertical transmission of HIV is independent of the length of time of rupture of membranes (as a secondary measure)

SECONDARY OUTCOMES:
Median length of time of membrane rupture | Ten Years
  In optimally managed HIV+ women with undetectable viral loads and on HAART, receiving intrapartum IV ZDV, the risk of vertical transmission of HIV is independent of the length of time of rupture of membranes (as a secondary measure)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yudin, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada